CLINICAL TRIAL: NCT05487716
Title: Effects of High-Intensity Interval Training on Long-term Survival in Patients With Different Heart Failure Phenotypes
Brief Title: HIIT Effects on Long-term Survival in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202200856B0
Record Dates: First submitted 2022-07-21; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-07

CONDITIONS: Morality; Remodeling, Ventricular; Heart Failure
Keywords: Aerobic exercise; Heart failure; Cardiac remodeling; Survival
MeSH Terms: conditions — Ventricular Remodeling; Heart Failure | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart failure patients (HF): Subjects in HF were subgrouped according to their baseline left ventricular ejection fraction obtained by 2-D echocardiography as HFrEF (LVEF<40%), HFmrEF (LVEF>=40% and <50%), and HFpEF (LVEF>50%)
  Subjects underwent an additional 36 sessions of high-intensity interval training (alternating 80% and 40% peak oxygen consumption) were considered HIIT participants in each subgroup (HFrEF, HFmrEF, HFpEF). Others without exercise intervention were considered multidisciplinary disease management program (MDP) participants.
  Interventions: Behavioral: High-intensity interval training (HIIT)

INTERVENTIONS:
Behavioral: High-intensity interval training (HIIT) — Included subjects who underwent an additional 36 sessions (2-3 sessions per week) of supervised bicycle ergometer (Ergoselect 150P, ergoline GmbH, Germany) training as in the previous protocol5 were classified as the HIIT participant. They exercised alternatively at 3-min interval of 80% VO2peak and 3-min interval of 40% VO2peak for 30 min each session.

SUMMARY:
The American Heart Association announces that exercise training should be considered for all stable cardiac patients (Class I, Level A). Therefore, exercise is an important issue for cardiac patients. It has also been reported that high-intensity interval training (HIIT) brings benefits on reversal of cardiac remodeling and long-term survival for HF patients. This study explores high-intensity interval training (HIIT) effects on long-term survivals in heart failure (HF) patients, diagnosed according to the Framingham criteria.

This retrospective cohort study is going to analyze HF patients diagnosed between January 1, 2009 and May 31, 2022 in a tertiary care hospital. All HF patients underwent the multidisciplinary disease management program (MDP) in the hospital were initially surveyed. Participants were further categorized into HF with reduced ejection fraction (HFrEF) (left ventricle ejection fraction [LVEF]<40%), HF with mildly reduced EF (HFmrEF) (LVEF>=40% and LVEF< 50%), and HF with preserved EF (HFpEF) ( LVEF>=50%) based on the initial 2-D echocardiography. Participants will be further divided into HIIT+MDP or MDP only in each group based on patient preference.

Age, sex, body height, body weight, disease duration, etiology for HF, co-morbidities, and medication were documented during follow-up (F/U). B-type natriuretic peptide, natriuretic peptide (BNP), cardiopulmonary exercise test (CPET) for peak oxygen consumption (VO2peak) and 2-D echocardiography for LV geometry were repeatedly assessed during follow-up. The end-point is the death of the patients or the date of May 31, 2022. All mortality causes and overall survival rates will be determined at the end of F/U.

HIIT effects on long-term survival (Kaplan-Meier survival curve) for patients with different heart failure phenotypes will be estimated by log rank test. Continuous variables between different groups were analyzed by student t-test, while continuous variables before and after HIIT within groups were assessed by paired t-test. Other non-continuous variables such as sex, and co-morbidities were compared by chi-square test.

DETAILED DESCRIPTION:
METHODS Participants The institutional review board of a tertiary care hospital approved the retrospective cohort study protocol. Patients with cardiovascular events between 1 January 2009 and 31 May 2022 in a tertiary care hospital and the following criteria were included.

* Patients with a diagnosis of HF according to the Framingham HF diagnostic criteria.
* HF patients with stable clinical presentation for> 4 weeks.

All included subjects received individualized patient education under optimized guideline-based management, i.e., multi-disciplinary disease management program (MDP), by the HF care team. Investigators excluded individuals based on the following criteria

* Age < 20 years and > 80 years.
* Pregnancy.
* Chance of cardiac transplantation within 6 months
* Moderate to severe chronic obstructive pulmonary disease
* Uncompensated HF.
* Estimated glomerular filtration rate < 30 ml/min/1.73m2
* Absolute contraindications for exercise suggested by the American College of Sports Medicine.
* Unable to perform exercise caused by non-cardiac disease.

Clinical Assessment Investigators recorded baseline age, sex, body mass index, co-morbidities, serum b-type natriuretic peptide levels, incremental cardiopulmonary exercise test (CPET) findings, and 2-D echocardiography measurements in all included participants. The physical component score (PCS) and mental component score (MCS) of the Medical Outcomes Study 36-item Short Form were used to evaluate quality of life (QoL) before initiating CPET.

Exercise Training Eligible HF patients who underwent an additional 36 sessions (2-3 sessions per week) of supervised bicycle ergometer (Ergoselect 150P, ergoline GmbH, Germany) training for 3-4 months were classified as the HIIT participant. Participants exercised alternatively at 3-min interval of 80% VO2peak and 3-min interval of 40% VO2peak for 30 min each session. The remaining participants without supervised HIIT were classified as the MDP participant.

Cardiopulmonary Exercise Test All participants underwent incremental CPET within 1 week before HIIT. Minute ventilation (VE) as well as CO2 ventilation (VCO2) and oxygen consumption (VO2) were measured breath by breath. VO2peak, VE-VCO2 slope, systemic arteriovenous O2 difference (Da-vO2), and peak cardiac output during the exercise test (COex) were defined.

Echocardiography 2-D echocardiography images were acquired at end-expiration with a 2-5 MHz tightly curved-array ultrasound transducer (Vivid 7, General Electric Healthcare, Chicago, IL, USA or Phillips IE33, Philips Healthcare, Andover, MA, USA) to measure LV end-diastolic dimension (LVEDD), LV end-systolic diameter (LVESD), and LVEF for all participants. HF patients with LVEF<40%, LVEF>= 40% and < 50%, and LVEF>=50% were considered to have HFrEF, HFmrEF, and HFpEF, respectively.

Follow-Up All participants were followed up until 31 May 2022 or when death occurred during the observational period. All HIIT participants underwent secondary CPET, QoL assessment, and 2-D echocardiography within 1 week after completing 36 sessions of HIIT. After completing the exercise training, HIIT participants received the same treatment program as the MDP participants until the end of F/U. 2-D echocardiography was performed during the long-term F/U at an interval of 3 to 12 months for all participants. Dates and causes of death were also documented.

Statistical Analysis Baseline demographic information between the HIIT and MDP participants with different HF phenotypes will be compared by Student's t test for continuous variables, and chi-squared test for categorical variables. For HIIT participants, ANOVA will be used to estimate differences in cardiorespiratory fitness and cardiac geometry after exercise training among the three phenotypes. Differences of the above evaluations between two among the three phenotypes will be estimated by the Bonferroni post hoc test. Paired t test will be used to assess HIIT effects on cardiorespiratory fitness and cardiac geometry in each phenotype.

To avoid immortal time bias, the index date for HIIT participants will be the date of exercise completion, while the index date for MDP participants will be the date of CPET examination. Kaplan-Meier survival curves for HF patients based on their exercise status for all HF patients and the different HF phenotypes will be assessed by log-rank test. The multivariable Cox regression will be used to investigate clinical predictors for mortality after conducting data exploration to select variables in the multivariable Cox model.

Heatmaps will be used to present the effect of HIIT on changes in LVEF and LV dimensions for different phenotypes during the long-term F/U. The HIIT-induced changes of LV geometry in each phenotype will be compared by Student's t test. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of heart failure according to the Framingham HF diagnostic criteria
* Stable heart failure clinical presentation for > 4 weeks.

Exclusion Criteria:

* Pregnancy
* Chance of cardiac transplantation within 6 months
* Moderate to severe chronic obstructive pulmonary disease
* Uncompensated heart failure
* Estimated glomerular filtration rate < 30 ml/min/1.73m^2
* Absolute contraindications for exercise suggested by the American College of Sports Medicine
* Unable to perform exercise caused by non-cardiac disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Included subjects with divided into three subgroups
  * Heart failure with reduced ejection fraction (HFrEF): LVEF <40%.
  * Heart failure with mildly reduced ejection fraction (HFmrEF): LVEF>=40% and < 50%.
  * Heart failure with preserved ejection fraction (HFpEF): LVELVEF>=50%.
  Among each group
  * High-intensity interval training (HIIT) participants: Included subjects who underwent 36 sessions (2-3 sessions per week) of hospital-based supervised bicycle ergometer training with alternatively at 3-min interval of 80% VO2peak and 3-min interval of 40% VO2peak for 30 min each session for 3-4 months
  * Multidisciplinary disease managment program (MDP) participants: Included subjects without hospital-based HIIT.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Death registration on our chart

SECONDARY OUTCOMES:
VO2peak in MET | From date of inclusion until 12-16 weeks after inclusion date
  Peak oxygen consumption
VE-VCO2 slope in (mL/min)/(mL/min) | From date of inclusion until 12-16 weeks after inclusion date
  Minute ventilation to CO2 production slope during cardiopulmonary exercise training
LVEF in % | through study completion, up to 12 years
  Left ventricular ejection fraction obtained from 2-D echocardiography
LVEDD in mm | through study completion, up to 12 years
  Left ventricular end-diastolic dimension obtained from 2-D echocardiography
LVESD in mm | through study completion, up to 12 years
  Left ventricular end-systolic dimension obtained from 2-D echocardiography
COex in mL/min | From date of inclusion until 12-16 weeks after inclusion date
  Peak cardiac output measured by the non-invasive cardiac output measurement during cardiopulmonary exercise test.
Da-vO2 in mL/dL | From date of inclusion until 12-16 weeks after inclusion date
  Systemic arteriovenous oxgen difference derived from VO2peak/COex

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chin Hsu, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chih-Chin Hsu, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
To assess the left ventricle (LV) remodeling response and long-term survival after high-intensity interval training (HIIT) in patients with various heart failure (HF) phenotypes.